CLINICAL TRIAL: NCT02064166
Title: A Double-blinded Placebo-controlled Single-center Study to Evaluate the Efficacy of Intranasal Insulin 40 International Units Day as Treatment for Subjects With Parkinson Disease and Multiple System Atrophy
Brief Title: Treatment of Parkinson Disease and Multiple System Atrophy Using Intranasal Insulin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Novak (Other)
Responsible Party: Sponsor-Investigator, Peter Novak, Former Faculty member, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PN-1
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease; Multiple System Atrophy
Keywords: Parkinson disease; Multiple system atrophy; Intranasal; Insulin
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin (Experimental): 40 IU of intranasal insulin daily
  Interventions: Drug: Intranasal Insulin
- Placebo (Placebo Comparator): Placebo arm using intranasal normal saline
  Interventions: Drug: Intranasal Insulin

INTERVENTIONS:
Drug: Intranasal Insulin — 1. treatment arm: Insulin, 40 international units daily, intranasally, for 4 weeks;
  2. placebo arm: normal saline, daily, intranasally, for 4 weeks.
  Other Names: Novolin R

SUMMARY:
Parkinson disease (PD) and multiple system atrophy (MSA) are progressive neurodegenerative disorders characterized by abnormal accumulation of α-synuclein. There is no effective treatment that can slow down the disease progression and both disorders are associated with severe cognitive decline. It was shown that intranasal insulin (INI) improves learning and memory in healthy and cognitively impaired non-diabetic adults.

The proof-of-concept, randomized, placebo-controlled, cross-over pilot study ( NCT01206322) has shown that a single 40 international units dose of intranasal insulin improves visuospatial memory in diabetes and control subjects.

This proposal includes randomized, double blinded, placebo-controlled trial of intranasal insulin (40 international units daily) in treatment of PD and MSA.

The study will evaluate 22 patients with PD and 22 patients with MSA. Total duration of the study will be 2 years. The primary goal is to assess the efficacy of INI in treatment of cognitive abnormalities in both PD and MSA. The primary efficacy end point will be change of the cognitive scale ratings.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females older than 17 years.
2. Clinical diagnosis of Parkinson disease or multiple system atrophy.
3. Provide written informed consent to participate in the study.
4. Understand that they may withdraw their consent at any time.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. In the investigator's opinion, have significant systemic, hepatic, cardiovascular, renal or other illness that can interfere based on investigator judgment with the trial.
3. History of dementia.
4. Unable to walk without help for at least 1 minute.
5. History of allergic reaction to insulin.
6. The presence of inflammation of nasal cavity that may prevents absorption of insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Novak', MD,PhD, Principal Investigator — Former Associate Professor
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Novak P, Pimentel Maldonado DA, Novak V. Safety and preliminary efficacy of intranasal insulin for cognitive impairment in Parkinson disease and multiple system atrophy: A double-blinded placebo-controlled pilot study. PLoS One. 2019 Apr 25;14(4):e0214364. doi: 10.1371/journal.pone.0214364. eCollection 2019. PMID 31022213

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin: Treatment arm: 40 IU of intranasal human insulin Novolin R, Novo Nordisk daily
  Intranasal Insulin: Insulin, 40 IU of daily, intranasally, for 4 weeks;
- Placebo: Placebo arm using intranasal normal saline
  Placebo arm: normal saline, daily, intranasally, for 4 weeks.
Period: Overall Study
Arm/Group | Insulin | Placebo
Started | 9 | 6
Completed | 8 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Insulin: 40 IU of intranasal insulin daily
  Intranasal Insulin: 1.treatment arm: Insulin, 40 international units daily, intranasally, for 4 weeks; 2. placebo arm: normal saline, daily, intranasally, for 4 weeks.
- Placebo: Placebo arm using intranasal normal saline
  Intranasal Insulin: 1.treatment arm: Insulin, 40 international units daily, intranasally, for 4 weeks; 2. placebo arm: normal saline, daily, intranasally, for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Insulin | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (5.7) | 62.2 (9.6) | 62.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Verbal Fluency FAS (F, A or S Words) Total Score
Description: Changes in Verbal Fluency FAS (a total number of F, A or S words) generated after 4 weeks of treatment compared to baseline, FAS total score is a sum of F,A, and S raw scores. The verbal fluency FAS test is used to assess phonemic fluency and verbal memory. Participants are asked to name words starting with letters F, A and S over one minute interval. The unit is a on scale, the normative data are adjusted for age and sex. The higher score means better verbal fluency.
Time Frame: Baseline and post-treatment
Measure: Mean (Standard Deviation); unit: Words
Groups:
- Insulin Baseline: FAS score in the insulin group at baseline Treatment arm: 40 IU of intranasal human insulin Novolin R, Novo Nordisk daily Intranasal Insulin: Insulin, 40 IU of daily, intranasally, for 4 weeks;
- Insulin Post Treatment: FAS score in the insulin group post treatment
  Treatment arm: 40 IU of intranasal human insulin Novolin R, Novo Nordisk daily Intranasal Insulin: Insulin, 40 IU of daily, intranasally, for 4 weeks;
- Placebo Baseline: FAS score in the placebo group at baseline Placebo arm using intranasal normal saline
  Placebo arm: normal saline, daily, intranasally, for 4 weeks.
- Placebo Post Treatment: FAS score in the placebo group post treatment Placebo arm using intranasal normal saline Placebo arm: normal saline, daily, intranasally, for 4 weeks
Arm/Group | Insulin Baseline | Insulin Post Treatment | Placebo Baseline | Placebo Post Treatment
Number analyzed (Participants) | 8 | 8 | 6 | 6
Words | 38.8 (5.7) | 41.0 (8.2) | 32.8 (2.3) | 30.8 (7.1)

2. Secondary Outcome: Modified Hoehn and Yahr Scale
Description: The modified Hoehn and Yahr Scale (HY) is used to assess severity of Parkinson Disease and treatment response post treatment as compared to baseline. The scale ranges from 1 to 5. The lower score indicates better outcome, e.g. less severe parkinsonism.
Time Frame: Baseline and post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Insulin Baseline: HY Scale in the insulin group at baseline
- Insulin Post Treatment: HY scale in the insulin group post treatment
- Placebo Baseline: HY scale in placebo group at baseline
- Placebo Post Treatment: HY scale in placebo group post treatment
Arm/Group | Insulin Baseline | Insulin Post Treatment | Placebo Baseline | Placebo Post Treatment
Number analyzed (Participants) | 8 | 8 | 6 | 6
score on a scale | 2.0 (0.6) | 2.0 (0.7) | 2.4 (0.38) | 2.4 (0.2)

3. Secondary Outcome: Cognitive Impairment Using Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) is a one-page 30-point test administered in approximately 10 minutes and is used to assess symptoms of cognitive impairment and their changes after treatment as compared to baseline. MoCA scores range between 0 and 30 with higher scores indicative of better cognitive performance. A score of 26 and above is considered to be normal.
Time Frame: Baseline and post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Insulin Baseline: MOCA Scale in insulin group at baseline
- Insulin Post Treatment: MOCA scale in insulin group post treatment
- Placebo Baseline: MOCA score in the placebo group at baseline
- Placebo Post Treatment: MOCA score in the placebo group post treatment
Arm/Group | Insulin Baseline | Insulin Post Treatment | Placebo Baseline | Placebo Post Treatment
Number analyzed (Participants) | 8 | 8 | 6 | 6
score on a scale | 28.7 (1.2) | 28.0 (1.1) | 26.8 (2.6) | 28.2 (0.95)

4. Secondary Outcome: Beck Depression Inventory Score (BDI)
Description: Beck Depression Inventory (BDI) is a 21-items self reported inventory with a scale evaluating depressive symptoms and the changes in BDI after treatment compared to baseline. The range of scores is 0 to 63, with higher scores indicating greater severity of depression.
Time Frame: Baseline and post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Insulin Baseline: BDI Scale in the insulin group at baseline
- Insulin Post Treatment: BDI scale in the insulin group post-treatment
- Placebo Baseline: BDI score in the placebo group at baseline
- Placebo Post Treatment: BDI score in the placebo group post treatment
Arm/Group | Insulin Baseline | Insulin Post Treatment | Placebo Baseline | Placebo Post Treatment
Number analyzed (Participants) | 8 | 8 | 6 | 6
score on a scale | 7.8 (5.4) | 8.25 (8.1) | 13.5 (5.6) | 12.8 (7.4)

5. Other Pre Specified Outcome: Unified Parkinson's Disease Rating Scale Part III (UPDRS Part III)
Description: UPDRS Part III has 14 items assessing motor skills including facial expression and speech, tremors, rigidity, posture, gait, and bradykinesia. Left and right sides (arms, legs, and hands) are assessed separately for seven of the functions. The total score for subscale 3 ranges from 0 to 108 (the sum of scores from 14 items with 27 observations). The higher the value, the more severe the symptoms. The outcomes reflect the UPDRS Part III score at baseline and 4 weeks post treatment with post treatment scores compared to baseline in the insulin and placebo groups.
Time Frame: Baseline and post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Insulin Baseline: UPDRS III Scale in the insulin group at baseline
- Insulin Post Treatment: UPDRS III Scale in the insulin group at post treatment
- Placebo Baseline: UPDRS III Scale in the placebo group at baseline
- Placebo Post Treatment: UPDRS III Scale in the insulin group post treatment
Arm/Group | Insulin Baseline | Insulin Post Treatment | Placebo Baseline | Placebo Post Treatment
Number analyzed (Participants) | 8 | 8 | 6 | 6
score on a scale | 31.5 (20.0) | 25.6 (21.8) | 31.7 (13.3) | 30.5 (15.8)

6. Other Pre Specified Outcome: Gait Analysis (4-meter Test)
Description: Changes in gait compared to baseline. Data are reported as changes in average stride interval ( inch) at baseline and post treatment.
Time Frame: Baseline and post-treatment
Measure: Mean (Standard Deviation); unit: inch
Groups:
- Insulin Baseline: Stride interval in the insulin group at baseline
- Insulin Post Treatment: Stride interval in the insulin group post treatment
- Placebo Baseline: Stride interval in placebo group at baseline
- Placebo Post Treatment: Stride interval in placebo group post treatment
Arm/Group | Insulin Baseline | Insulin Post Treatment | Placebo Baseline | Placebo Post Treatment
Number analyzed (Participants) | 8 | 8 | 6 | 6
inch | 22.0 (5.0) | 21.5 (4.4) | 21.0 (2.7) | 19.6 (2.9)

7. Other Pre Specified Outcome: Brief Visuospatial Memory Test-Revised (BVMT-R)
Description: Changes in Brief Visuospatial Memory Test-Revised (BMVT-R) compared to baseline. For BVMT, there were concerns about the test administration and validity of this test which relies on fine motor control in PD patients that have motor impairment which could affect the drawing precision. Therefore, BVMT was not included in the analyses, because these methodological concerns would have affected the calculation of the total score as the outcome measure.
Time Frame: Baseline and post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Insulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 1/9 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin (N=9) | Placebo (N=6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No